CLINICAL TRIAL: NCT02057302
Title: A Multicenter, Pragmatic Randomized, Double-blind, Placebo-controlled Trial of Xuezhikang Capsule for Treating Dyslipidemia: a Postmarketing Study
Brief Title: A Study on Postmarketing Xuezhikang Capsule for Treating Dyslipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Xing Liao, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008ZX09202-007
Record Dates: First submitted 2014-01-28; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Dyslipidemia
Keywords: Xuezhikang Dyslipidemia chinese medicine RCT
MeSH Terms: conditions — Dyslipidemias | interventions — xuezhikang

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Placebo Comparator): There are 538 patients recruited in this group. Patients in this group will take 2 capsules of placebo every time, twice every day, respectively after breakfast and supper.
- Group A (Experimental): There are 1614 patients recruited in this group. Patients in this group will take 2 capsules of Xuezhikang every time, twice every day, respectively after breakfast and supper.
  Interventions: Drug: Xuezhikang capsule

INTERVENTIONS:
Drug: Xuezhikang capsule
  Arms: Group A

SUMMARY:
Dyslipidemia contributes greatly to the formation and progression of atherosclerosis (AS), which plays a dominant role in leading to CHD.

Xuezhikang is a partially purified extract of fermented red yeast rice (Monascus purpureus). It is composed of 13 kinds of natural statins, unsaturated fatty acids, ergosterol,amino acids, flavonoids, alkaloid, trace element, and so forth. Xuezhikang has been recommended in a guideline for China adult dyslipidemia prevention.

This study aims to evaluate the benefit and side effect of Xuezhikang, a potential alternative drug of statins, for patients with dyslipidemia, and thus provide further evidence for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years to 75 years
2. Patients with Dyslipidemia should be diagnosed according to standard western medicine diagnosis criteria
3. TCM syndrome of patients with dyslipidemia should be diagnosed according to standard TCM syndrome diagnosis criteria
4. Patients who have taken lipid lowering drugs should stop taking for at least two weeks before taking part in this study
5. Patients agree to participate in this study and signed the informed consent form

Exclusion Criteria:

1. Pregnant (positive pregnancy test within 7 days of starting treatment), or lactating women.
2. Patients with Homozygous Familial Hypercholesterolemia
3. Patients with known allergy to Chinese medicine or any other drug
4. Patients with acute myocardial infarction, cerebrovascular accident , severe trauma , major surgery and cancer in half a year.
5. AST or ALT level increases at least twice the upper limits of normal in patients
6. Patients who are taking part in other clinical trials that will influence the results of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Blood samples were drawn were detected,including TC,TG,LDL-C and HDL-C | the detect the change from baseline to the 8th week

SECONDARY OUTCOMES:
Traditional Chinese medicine syndrome scores (TCM-SS) and single TCM symptom | to detect the change at baseline, 2nd week, 4th week, 6th week, and 8th week

OTHER OUTCOMES:
safety outcomes including vital signs and laboratory tests | to detect the change from baseline to 8th week